CLINICAL TRIAL: NCT07019480
Title: Influence of Implant Insertion Torque on Post-Surgical Marginal Bone Stability: A Multicenter Clinical Study
Brief Title: Influence of Implant Insertion Torque on Post-Surgical Marginal Bone Stability
Status: Active, not recruiting | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Sponsor
Other Study IDs: MEGAWH 1.0
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort: implant insertion with recorded torque and stability values
  Interventions: Procedure: implant insertion

INTERVENTIONS:
Procedure: implant insertion — Following local anesthesia (articaine 4% with epinephrine 1:100,000), a minimally invasive full-thickness flap will be elevated. Implant site preparation will be performed with twist drills and the implant will be inserted. Implant stability (ISQ) will be measured in the mesio-distal, disto-mesial, bucco-lingual, and linguo-buccal directions using a resonance frequency analysis device (Osstell Beacon, Osstell, Göteborg, Sweden) with a single-use magnetic peg specific to the implant (SmartPeg Type 07, Osstell, Göteborg, Sweden).
  The flap will be closed using non-resorbable monofilament sutures, and the implant will be submerged (two-stage protocol).

SUMMARY:
The aim of this prospective, multicenter observational study is to evaluate the influence of various surgical parameters (maximum insertion torque; average insertion torque; final insertion torque; area under the torque curve; intercept and slope of the least squares regression line of the torque curve; implant stability quotient measured immediately after implant insertion) on implant osseointegration and on peri-implant marginal bone loss occurring during the first three months of submerged healing.

DETAILED DESCRIPTION:
This proposed study is a prospective, observational multicenter clinical trial. Ten independent clinical centers will treat partially edentulous patients with dental implants following a specific surgical protocol.

Enrollment Procedure: All patients meeting the inclusion and exclusion criteria will be enrolled in the study after receiving the Information Sheet and providing written informed consent.

Pre-surgical planning will be performed using a CBCT scan with or without the aid of dedicated image reconstruction software. A preoperative periapical radiograph will also be taken using a customized Rinn-type film holder for each patient, with the aid of a silicone key.

Surgical phase: After local anesthesia with 4% articaine containing 1:100,000 epinephrine, a minimally invasive full-thickness mucoperiosteal flap will be elevated to visualize the crest anatomy. The height of the supracrestal soft tissue will be measured using a dedicated probe (SSL, Medesy, Maniago, Italy) and categorized as thin (<2.5 mm), medium (2.5-3.5 mm), or thick (>3.5 mm).

Implant site preparation will be carried out using a dedicated surgical kit (Anyone, Megagen, Gyeongbuk, South Korea). The implant (Anyone, 4.0×8.5 mm) will then be placed at crestal level, with torque values recorded throughout the entire insertion process using a surgical motor set to 30 rpm (Implantmed, W&H, Burmoos, Austria). The maximum torque will be limited to 80 Ncm.

If the maximum torque is insufficient to complete insertion, the implant will be removed and the site will be further prepared using the next drill in the sequence.

After crestal-level placement, Patients will be prescribed an NSAID (ibuprofimplant stability (ISQ) will be measured in the mesio-distal, disto-mesial, bucco-lingual, and linguo-buccal directions using a resonance frequency analysis device (Osstell Beacon, Osstell, Göteborg, Sweden) with a single-use magnetic peg specific to the implant (SmartPeg Type 07, Osstell, Göteborg, Sweden). Calibration of the device must be verified prior to each patient procedure using an implant secured in a resin block.

The flap will be closed using non-resorbable monofilament sutures, and the implant will be submerged (two-stage protocol). A periapical radiograph will be taken at this point (T0) using the previously described customized Rinn-type holder. en 600 mg, as needed) and instructed to rinse with 0.2% chlorhexidine mouthwash for two minutes, three times per day, starting on the second postoperative day.

Sutures will be removed 7-10 days after surgery.

Post-surgical follow-ups: After three months of healing (T1), a periapical radiograph will be taken using the previously described customized holder, and a second-stage surgery will be performed to uncover the implant. Following ISQ measurement as previously described, a definitive transmucosal abutment of appropriate length and diameter (OCTA, Megagen, Gyeongbuk, South Korea) will be connected. After a four-week healing period, an abutment-level impression will be taken for the fabrication of the final prosthesis, which may be either a single screw-retained metal-ceramic crown or a screw-retained bridge.

Periapical radiographic follow-ups will be performed as described above at prosthesis delivery and at 6 months, 1 year, 3 years, and 5 years post-loading to assess marginal bone stability.

Radiographic Measurements: All radiographs will be taken using identical radiographic device settings (60 kV, 7 mA). Peri-implant bone levels (PBL) will be measured at T0 and T1 as the linear distance between the implant platform and the bone crest at the mesial and distal aspects of each implant. A positive value will be assigned when the bone crest is coronal to the implant platform, while a negative value will be recorded when the first bone-to-implant contact is apical to the implant platform.

The difference in PBL between T0 and T1 will represent marginal bone loss if PBL_T1 < PBL_T0, and marginal bone gain if PBL_T1 > PBL_T0. Measurements will be calibrated according to the known implant diameter and length.

Any radiograph showing distortion and/or other quality issues must be immediately retaken.

All measurements will be performed by two blinded examiners using image analysis software (ImageJ 1.52a, National Institutes of Health, Bethesda, MD, USA) on a 24-inch medical-grade monitor. Each measurement will be repeated three times at three different time points, as proposed by Gomez-Roman and Launer.

Examiner calibration will be carried out on a sample of ten radiographs not included in the study. The Cohen's kappa coefficient (k) will be calculated by a third investigator to assess intra-examiner and inter-examiner agreement.

Statistical Analysis: Descriptive statistics will be used to summarize the baseline characteristics of the study population. The relationship between insertion torque and marginal bone loss will be assessed using regression models, adjusting for potential confounding variables. Repeated measures ANOVA will be used to analyze ISQ changes over time. A p-value <0.05 will be considered statistically significant. Data analysis will be performed using SPSS Statistics v25.0 (IBM Corp., Armonk, NY, USA).

Sample Size Calculation: The sample size was calculated based on a previously published study (Marconcini S, Longitudinal analysis on the effect of insertion torque on delayed single implants: A 3-year randomized clinical study. Clin Implant Dent Relat Res. 2018;20(3):322-332.), which reported a one-year failure rate of 1.72% (1/58) in the low insertion torque group (<50 Ncm) and 3.45% (2/58) in the high insertion torque group (≥ 50 Ncm). A 1:1 allocation ratio was considered, with a significance level of 0.01 and statistical power of 90%. The minimum required sample size was 68 implants (34 per group). To compensate for potential drop-outs and to allow for repeated measures analysis, 150 implants will be placed across 10 clinical centers (15 implants per center). Each patient may contribute up to 3 implants.

ELIGIBILITY:
Inclusion Criteria:

* Indication for implant-supported prosthetic rehabilitation of single or multiple partial edentulism in one or both arches, based on accurate diagnosis and treatment planning;
* The area in which the implants will be placed must have had at least 6 months of healing;
* Residual alveolar ridge width ≥7 mm;
* Available bone height >9 mm at the planned implant site;
* Patient aged >18 years;
* Patient does not use any removable prosthesis at the site to be treated;
* Patient is able and willing to comply with the study protocol;
* Patient signs the written informed consent.

Exclusion Criteria:

* Acute myocardial infarction within the past two months;
* Uncontrolled bleeding disorders;
* Uncontrolled diabetes (HBA1c > 7.5);
* History of head and/or neck radiotherapy within the past 24 months;
* Immunocompromised patients, HIV positive, or undergoing chemotherapy within the past five years;
* Current or previous antiresorptive therapy;
* Psychological or psychiatric disorders;
* Drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After investigating general and local anamnesis, which included evaluation of systemic illnesses and potential allergies, a dental visit was conducted to formulate a specific treatment plan.
  If the patient was deemed eligible for the research protocol, an additional periapical radiograph was obtained for each selected site to assess the adequacy of residual bone height.
  If the available bone height appeared to be sufficient, a second-level radiographic exam, a Cone Beam Computed Tomography (CBCT), was performed to evaluate whether the bone volume was adequate for supporting implant rehabilitation.
  For patients requiring tooth extraction, this second assessment was performed after six months of healing after extraction.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant Stability Quotient (ISQ) for the evaluation of primary stability, measured using a resonance frequency analysis (RFA) device (Osstell). | Immediately after implant placement
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden). ISQ will be measure in the mesio-distal, disto-mesial, bucco-lingual, and linguo-buccal directions.
Implant primary stability in Newton | During the full course of implant insertion
  Insertion torque
Periapical radiograph for the assessment of peri-implant bone level (PBL) in millimeters | Immediately after implant placement
  Periapical radiograph using a customized Rinn-type film holder for each patient with the aid of a silicone index

SECONDARY OUTCOMES:
Implant Stability Quotient (ISQ) for the evaluation of secondary stability, measured using a resonance frequency analysis (RFA) device (Osstell) | 3 months after implant insertion
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden). ISQ will be measure in the mesio-distal, disto-mesial, bucco-lingual, and linguo-buccal directions.
Periapical radiograph for the assessment of peri-implant bone level (PBL) in millimeters | 3 months after implant insertion
  Periapical radiograph using a customized Rinn-type film holder for each patient with the aid of a silicone index
Periapical radiograph for the assessment of peri-implant bone level (PBL) in millimeters | upon prosthesis delivery
  Periapical radiograph using a customized Rinn-type film holder for each patient with the aid of a silicone index
Periapical radiograph for the assessment of peri-implant bone level (PBL) in millimeters | 6 months after prosthetic loading
  Periapical radiograph using a customized Rinn-type film holder for each patient with the aid of a silicone index
Periapical radiograph for the assessment of peri-implant bone level (PBL) in millimeters | 1 year after prosthetic loading
  Periapical radiograph using a customized Rinn-type film holder for each patient with the aid of a silicone index
Periapical radiograph for the assessment of peri-implant bone level (PBL) in millimeters | 3 years after prosthetic loading
  Periapical radiograph using a customized Rinn-type film holder for each patient with the aid of a silicone index
Periapical radiograph for the assessment of peri-implant bone level (PBL) in millimeters | 5 years after prosthetic loading
  Periapical radiograph using a customized Rinn-type film holder for each patient with the aid of a silicone index

CONTACTS AND LOCATIONS:
Locations (1):
- University of Trieste, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: No